CLINICAL TRIAL: NCT06910007
Title: Accuracy of Advanced Treatment Planning Software for Static Computer Guided Surgery ( Blue Sky Plan Bio, Exoplan, Real Guide Computer Software)
Brief Title: Accuracy of Various Advanced Treatment Planning Software for Static Computer Guided Surgery in Dental Implant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hussein Anssari, PhD student in oral and maxillofacial surgery, University of Baghdad
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1025 in 11-2-2025
Record Dates: First submitted 2025-03-22; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Dental Implant
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- blue sky plan group (Active Comparator): surgical guide will be fabricated using Blue sky plan computer software
  Interventions: Procedure: dental implant will be inserted using surgical guide; Procedure: dental implant
- exoplan group (Active Comparator): surgical guide will be fabricated using Exoplan computer software
  Interventions: Procedure: dental implant will be inserted using surgical guide; Procedure: dental implant
- Real guide group (Active Comparator): surgical guide will be fabricated using Real guide computer software
  Interventions: Procedure: dental implant will be inserted using surgical guide; Procedure: dental implant

INTERVENTIONS:
Procedure: dental implant will be inserted using surgical guide — dental implant will be inserted using blue sky plan computer software
Procedure: dental implant — surgical guide will be fabricated using exoplan computer software
Procedure: dental implant will be inserted using surgical guide — surgical guide will be fabricated using real guide computer software

SUMMARY:
This study will be conducted to investigate the accuracy of Blue sky plan bio , exoplan ,and real guide advanced treatment planning software required for static computer guided surgery designing and manufacturing.

ELIGIBILITY:
Inclusion Criteria:

1. partially edentulous adults with at least three teeth remaining.
2. an expected sufficient bone volume to perform implant insertion with at least a 3.5mm Cybermed dental implant without simultaneous bone augmentation.
3. extractions performed at least 3 months earlier.
4. potential earlier sinus grafting was performed at least 6 months prior to implant placement.
5. Patients with absence of any periodontal problems in the adjacent teeth.

7- stable medical condition to undergo implant surgery (ASA 1 or 2).

Exclusion Criteria:

1. Physical or psychological disorders generally prohibiting implant therapy. After initial screening.
2. Patients with a history of bruxism
3. Patients with over eruption of the opposing tooth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2026-11-28 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
deviation between planned and actual implant position when using different planning software | 14 days
  measurement will be done by superimposition two CBCTs showing the pre-operation ( planned) and post operation implant position which will reveal the deviation in millimeter in regards to entry point ,apical ,and angular deviation of dental implant using specified tool within the planning software

IPD SHARING:
Plan to Share IPD: No